CLINICAL TRIAL: NCT00367601
Title: A Phase II Study of Erlotinib With Bevacizumab in Chemotherapy Naïve Performance Status (PS) 2 Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: Erlotinib + Bevacizumab for PS 2 Chemotherapy Naïve Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nasser Hanna, M.D. (Other)
Collaborators: Genentech, Inc. (Industry); Walther Cancer Institute (Other); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Nasser Hanna, M.D., Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LUN04-77
Record Dates: First submitted 2006-08-21; First posted 2006-08-23 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Erlotinib Hydrochloride; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Bevacizumab + erlotinib; if no progressive disease observed, combination or single-agent treatment will continue until unacceptable toxicity or progressive disease.
  Interventions: Drug: Erlotinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg qd days 1-21
Drug: Bevacizumab — Bevacizumab 15 mg/kg IV, day 1

SUMMARY:
The strategy for combining therapeutic agents in cancer treatments has been successful in multiple tumor types, including NSCLC. Erlotinib and bevacizumab target different pathways involved in tumor growth. Nonclinical studies have demonstrated that the combination of bevacizumab and erlotinib results in greater efficacy than either agent alone. Furthermore, because there is little to no overlap in toxicity profile between the two agents, the combination is expected to be well tolerated and may provide even greater benefit for patients who are unable to receive cytotoxic therapy.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Bevacizumab 15 mg/kg IV on day 1
* Erlotinib 150 mg po qd days 1-21
* Disease Assessment during even numbered cycles

If no progressive disease observed, continue (combination or single agent- see below) until unacceptable toxicity or progressive disease.

If progressive disease observed, treatment will be discontinued.

* Cycles will be repeated every 21 days up to a total of 6 cycles.
* Patients with non-progression after 6 cycles may stay on therapy (single agent erlotinib or the combination) until progressive disease or intolerable toxicity (at the physician discretion).
* Patients who require discontinuation of bevacizumab may receive at investigator's discretion erlotinib alone on study until progression.
* Patients who require discontinuation of erlotinib may receive at investigator's discretion bevacizumab alone until progression.

ECOG Performance Status 2

Hematopoietic:

* Absolute neutrophil count (ANC) > 1,000 mm3
* Platelet count > 100,000 mm3
* Hemoglobin > 8 g/dl

Hepatic:

* Bilirubin < 2 X upper limit of normal.
* Aspartate aminotransferase (AST, SGOT) < 2.5 X upper limit of normal or 5 X if liver involvement.

Renal:

* Urine protein:creatinine ratio 1.0 at screening

Cardiovascular:

* Blood pressure of < 150/100 mmHg.
* No history of unstable angina.
* No history of New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* No history of myocardial infarction within 6 months prior to registration for protocol therapy.
* No history of stroke within 6 months prior to registration for protocol therapy.
* No clinically significant peripheral vascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Histological proof of non-small cell lung cancer meeting one of the following criteria:

  * stage III b with a pleural effusion
  * stage IV
* Histology must not be squamous cell.
* No prior chemotherapy or hormonal therapy.
* Prior radiation therapy must be completed at least 21 days prior to being registered for protocol therapy.
* No prior use of an epidermal growth factor receptor (EGFR) inhibitor or antiangiogenic agent.
* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
* Measurable disease according to RECIST and obtained by imaging within 28 days prior to being registered for protocol therapy.
* ECOG Performance Status of 2 in the opinion of the treating investigator.
* Age > 18 years at the time of consent.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) while on treatment and for a 6 week period thereafter.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy. Subjects are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Females must not be breastfeeding.
* Able to comply with study and/or follow-up procedures.

Exclusion Criteria:

* Evidence of bleeding diathesis or coagulopathy.
* Evidence of central nervous system involvement or brain metastases confirmed by head CT or brain MRI within 28 days prior to being registered for protocol therapy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration for protocol therapy.
* Anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to registration for protocol therapy.
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to registration for protocol therapy.
* Serious, non-healing wound, ulcer, or bone fracture.
* History of hemoptysis.
* Clinically significant infections as judged by the treating investigator.
* Other active malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-08; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (13):
- United States (13):
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Methodist Cancer Center, Omaha, Nebraska
  - Oncology Partners Network, Cincinnati, Ohio

REFERENCES:
- [Result] T. Al Baghdadi, S. Bhatia, W. Harb, J. Maher, J. McClean, S. Nattam, D. Taber, M. Yu, C. Johnson and N. Hanna. Erlotinib and bevacizumab in chemotherapy naïve performance status 2 patients with advanced non-small-cell lung cancer. Accepted (abstract #e19082) at the ASCO annual meeting May 29-June 2, 2009, Orlando, FL
- [Result] Riggs H, Jalal SI, Baghdadi TA, Bhatia S, McClean J, Johnson C, Yu M, Taber D, Harb W, Hanna N. Erlotinib and bevacizumab in newly diagnosed performance status 2 or elderly patients with nonsquamous non-small-cell lung cancer, a phase II study of the Hoosier Oncology Group: LUN04-77. Clin Lung Cancer. 2013 May;14(3):224-9. doi: 10.1016/j.cllc.2012.09.004. Epub 2012 Oct 24. PMID 23102811
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Assignment: Bevacizumab + erlotinib; if no progressive disease observed, combination or single-agent treatment will continue until unacceptable toxicity or progressive disease.
  Erlotinib: Erlotinib 150 mg qd days 1-21
  Bevacizumab: Bevacizumab 15 mg/kg IV, day 1
Period: Overall Study
Arm/Group | Single Arm Assignment
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 25
Age, Customized [Median (Full Range); unit: years]
  Median Age, Years | 77 [52 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Investigator Assigned Performance Status [Number; unit: participants]
  Performance Status 1 | 2
  Performance Status 2 | 23
Patient-Reported Performance Status [Number; unit: participants]
  Performance Status 1 | 8
  Performance Status 2 | 13
  Performance Status 3 | 2
  Performance Status Missing | 2
Smoking Status [Number; unit: participants]
  Never Smoked | 1
  Not smoked in > 30 years | 4
  Quit > 3 months ago but <30 years ago | 10
  Current smoker | 9
  Unknown | 1
Stage [Number; unit: participants]
  Stage III-B | 3
  Stage IV | 22

OUTCOME MEASURES:

1. Primary Outcome: To Establish Rate of Non-progressive Disease at 4 Months in Patients With Advanced NSCLC Who Have Been Designated PS2 by Their Treating Physician
Time Frame: 4 months
Measure: Number; unit: percentage of participants
Groups:
- Single Arm: Bevacizumab + erlotinib; if no progressive disease observed, combination or single-agent treatment will continue until unacceptable toxicity or progressive disease.
Arm/Group | Single Arm
Number analyzed (Participants) | 25
percentage of participants | 28

2. Secondary Outcome: Time to Progression
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 25
months | 3.4 [1.3 to 5.4]

3. Secondary Outcome: Overall Survival
Time Frame: 12 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm Assignment
Number analyzed (Participants) | 25
months | 5.1 [3.3 to 8.3]

ADVERSE EVENTS:
Arm/Group | Single Arm Assignment
Serious Adverse Events (participants affected / at risk) | 16/25
Other Adverse Events (participants affected / at risk) | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Assignment (N=25)
ADULT RESPIRATORY DISTRESS SYNDROME (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 3 (3)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 1 (2)
FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (2)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
PAIN / BACK (General disorders) | 1 (1)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
ULCER, GI / DUODENUM (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Assignment (N=25)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 1 (1)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 11 (14)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
BRONCHOSPASM, WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1)
CARDIAC ARRHYTHMIA - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (7)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (11)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 11 (16)
DIZZINESS (Nervous system disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 7 (8)
EDEMA: LIMB (Blood and lymphatic system disorders) | 4 (4)
EXTREMITY-LOWER (GAIT/WALKING) (Musculoskeletal and connective tissue disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 11 (16)
FRACTURE (Musculoskeletal and connective tissue disorders) | 2 (2)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 3 (3)
HEMOGLOBIN (Blood and lymphatic system disorders) | 3 (3)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HYPOTENSION (Cardiac disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 3 (4)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / ABDOMEN NOS (Infections and infestations) | 2 (2)
INFECTION WITH UNKNOWN ANC / SKIN (CELLULITES) (Infections and infestations) | 2 (2)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 2 (3)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 2 (2)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 4 (4)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 4 (8)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 2 (2)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 6 (7)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 1 (1)
NEUROPATHY: MOTOR (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2)
OCULAR SURFACE DISEASE (Eye disorders) | 1 (1)
OCULAR/VISUAL - OTHER (SPECIFY, __) (Eye disorders) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / BACK (General disorders) | 1 (1)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / FACE (General disorders) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 1 (1)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / NECK (General disorders) | 1 (1)
PAIN / SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
PAIN / TUMOR PAIN (General disorders) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 1 (1)
PANCREATIC ENDOCRINE: GLUCOSE INTOLERANCE (Endocrine disorders) | 2 (2)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 3 (3)
PROTEINURIA (Investigations) | 4 (4)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 10 (19)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (3)
RASH: ERYTHEMA MULTIFORME (E.G., STEVENS-JOHNSON SYNDROME, TOXIC EPIDERMAL NECROLYSIS) (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN BREAKDOWN/DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (2)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 1 (1)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1)
VASCULAR - OTHER (SPECIFY, __) (Vascular disorders) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 2 (2)
WEIGHT GAIN (General disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 1 (1)
WOUND COMPLICATION, NON-INFECTIOUS (Skin and subcutaneous tissue disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No